CLINICAL TRIAL: NCT02656680
Title: Developing an Effective Online Social Network for Weight Loss
Brief Title: Facebook and Friends: Developing an Effective Online Social Network for Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Sherry Pagoto, Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H17-215; 1K24HL124366-01A1 (NIH)
Record Dates: First submitted 2016-01-07; First posted 2016-01-15 (Estimated); Results first posted 2021-03-16 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Continuous Enrollment (Randomized) (Experimental): The Continuous Enrollment is a Facebook-delivered weight loss intervention. Participants in this arm were randomized to this Facebook group and started the intervention together. For this group, the study team continued to enroll participants through week 8.
  Interventions: Behavioral: Continuous Enrollment
- Closed Enrollment (Randomized) (Active Comparator): Closed Enrollment is a Facebook-delivered weight loss intervention. Participants in this arm were randomized to this Facebook group and started the intervention together. No additional participants were added to this group during the study.
  Interventions: Behavioral: Closed Enrollment
- Continuous Enrollment (Non-Randomized) (Other): The Continuous Enrollment is a Facebook-delivered weight loss intervention. For this group, the study team continued to enroll participants through week 8. This arm captures only those participants that were added to the group during these 8 weeks. They were enrolled in the study after the original 80 participants were randomized.
  Interventions: Behavioral: Continuous Enrollment

INTERVENTIONS:
Behavioral: Continuous Enrollment — Participants will receive a weight loss intervention delivered in an online context. The online coaches will post daily content, respond to questions, address concerns, and encourage engagement. The weight loss intervention is based on the Diabetes Prevention Program (DPP), an evidence-based weight loss program focused on lifestyle changes. The goals for the intervention are 175 minutes of moderate physical activity per week and an overall weight loss of 7%. Each participant will get an individualized calorie goal that would facilitate a 1-2 lbs. weight loss weekly. Participants will also be encouraged to use an app such as MyFitnessPal to track daily diet. For this arm, the study team will keep recruitment open for this condition to allow enrollment of new participants through week 8.
  Other Names: Open Group
  Arms: Continuous Enrollment (Non-Randomized); Continuous Enrollment (Randomized)
Behavioral: Closed Enrollment — Participants will receive a weight loss intervention delivered in an online context. The online coaches will post daily content, respond to questions, address concerns, and encourage engagement. The weight loss intervention is based on the Diabetes Prevention Program (DPP), an evidence-based weight loss program focused on lifestyle changes. The goals for the intervention are 175 minutes of moderate physical activity per week and an overall weight loss of 7%. Each participant will get an individualized calorie goal that would facilitate a 1-2 lbs. weight loss weekly. Participants will also be encouraged to use an app such as MyFitnessPal to track daily diet.
  Other Names: Closed Group
  Arms: Closed Enrollment (Randomized)

SUMMARY:
In a pilot randomized trial of 160 obese participants, investigators will test the feasibility of a behavioral weight loss program delivered entirely via Facebook. We will recruit in 2 separate waves of 80 participants each. Participants will be randomized to: 1) a condition with study participants only or 2) to a condition they will be able to invite their friends into (wave 1) or one in which the study team keeps recruitment open to allow enrollment through week 8 (wave 2). All participants will receive behavioral counseling via the private Facebook group from the coaches who are present on the network daily. Participants will track their diet and exercise via a free commercial mobile app.

DETAILED DESCRIPTION:
The overarching goal of the research plan is to test ways to leverage mobile technologies and social media to increase the impact, scalability, cost-effectiveness, and dissemination potential of lifestyle interventions that reduce cardiovascular disease (CVD) risk. Mobile technology and social media have the potential to reduce the intensity of traditional prevention interventions and enhance outcome by delivering behavioral strategies in-the-moment and by connecting patients other patients to generate better communication and a social support system for lifestyle changes.

This study includes a behavioral weight loss program delivered entirely via on online social network. The weight loss intervention is based on the Diabetes Prevention Program (DPP), an evidence-based weight loss program focused on lifestyle changes. The goals for the intervention are 175 minutes of moderate physical activity per week and an overall weight loss of 7%. Each participant will get an individualized calorie goal that would facilitate a 1-2 lbs. weight loss weekly. Participants will be connected to one another via Facebook and receive behavioral counseling via posts from coaches who are present on the network daily. Participants will track their diet and exercise via a free commercial mobile app. Participants will be assigned to either a Facebook group allowing the invite of friends (wave 1), a Facebook group with open enrollment through week 8 (wave 2) or a Facebook group including only study participants. If they are assigned to the group including their friends, they have the opportunity to invite their friends to participate in the weight loss group if they are interested in losing weight as well. They will not have a limit as to how many friends they can invite. The friends that are invited will not undergo the same procedures as the Facebook (FB)+friends study participants, but we will provide them with a factsheet and collect minimal information from them. If they are assigned to the group with open enrollment through week 8, additional people will be recruited into that group. Those participants being enrolled between week 1-8 will undergo the same procedures as others besides randomization. The goal of both of these studies is to explore how to build the size of online weight loss groups in such a way that increases participant engagement. Feasibility outcomes include engagement (frequency of posts, likes, and comments and number of completed days of tracking posted) retention, acceptability, and weight loss. Post intervention focus groups will gather feedback on the program.

ELIGIBILITY:
Inclusion Criteria:

Participants must be:

1. 18-65 years of age;
2. Have a BMI 27-45 kg/m²;
3. Lives in the United States; and
4. Have daily internet access;

Exclusion Criteria:

1. Does not post on Facebook at least once per week
2. Comments on someone else's post on Facebook less than once per week
3. Does not currently use a smartphone;
4. Is not familiar with using phone apps;
5. Pregnant and/or lactating;
6. Meets criteria for severe depression on the Patient Health Questionnaire (PHQ-9) (score of >20);
7. Had bariatric surgery, plans to during the study;
8. Has had a weight loss of 5% or greater within previous 3 months;
9. Meets criteria for Binge Eating Disorder;
10. Condition that precludes lifestyle changes (i.e. a condition that prevents physical activity increase or dietary changes);
11. Medications affecting weight;
12. Incapable of walking ¼ mile without stopping;
13. Type 1 or 2 diabetes;
14. Participated in previous weight loss studies under the PI;
15. Has concerns about being in a Facebook group with other faculty, staff, or students from the University of Connecticut;
16. Has concerns about being audiotaped;
17. Inability to provide consent;
18. Prisoners; and
19. Non-English speaking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherry Pagoto, PhD, Principal Investigator — University of Connecticut
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu R, Divito J, Bannor R, Schroeder M, Pagoto S. Predicting Participant Engagement in a Social Media-Delivered Lifestyle Intervention Using Microlevel Conversational Data: Secondary Analysis of Data From a Pilot Randomized Controlled Trial. JMIR Form Res. 2022 Jul 28;6(7):e38068. doi: 10.2196/38068. PMID 35900824
- [Derived] Pagoto SL, Schroeder MW, Xu R, Waring ME, Groshon L, Goetz JM, Idiong C, Troy H, DiVito J, Bannor R. A Facebook-Delivered Weight Loss Intervention Using Open Enrollment: Randomized Pilot Feasibility Trial. JMIR Form Res. 2022 May 6;6(5):e33663. doi: 10.2196/33663. PMID 35522466

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: At the start of the 16-week trial, we randomized participants (n=80) to two groups: 'Facebook (FB)+Friends' (n=40) or 'FB Only' (n=40). For the first 8 weeks of the trial, we continued to add new participants (n=54) into the 'FB+Friends' group. Our total enrollment (n=134) includes these 54 post-randomized participants. We did not include the post-randomized sample in the analysis for this record.
Groups:
- FB+Friends: FB+Friends is a Facebook-delivered weight loss intervention. The study team will keep recruitment open for this condition to allow enrollment through week 8.
  Participants will receive a weight loss intervention delivered in an online context. The online coaches will post daily content, respond to questions, address concerns, and encourage engagement. The weight loss intervention is based on the Diabetes Prevention Program (DPP), an evidence-based weight loss program focused on lifestyle changes. The goals for the intervention are 175 minutes of moderate physical activity per week and an overall weight loss of 7%. Each participant will get an individualized calorie goal that would facilitate a 1-2 lbs. weight loss weekly. Participants will also be encouraged to use an app such as MyFitnessPal to track daily diet. For this arm, the study team will keep recruitment open for this condition to allow enrollment of new participants through week 8.
- FB Only: FB Only Facebook-delivered weight loss intervention including only study participants.
  FB Only: Participants will receive a weight loss intervention delivered in an online context. The online coaches will post daily content, respond to questions, address concerns, and encourage engagement. The weight loss intervention is based on the Diabetes Prevention Program (DPP), an evidence-based weight loss program focused on lifestyle changes. The goals for the intervention are 175 minutes of moderate physical activity per week and an overall weight loss of 7%. Each participant will get an individualized calorie goal that would facilitate a 1-2 lbs. weight loss weekly. Participants will also be encouraged to use an app such as MyFitnessPal to track daily diet.
- Non-Randomized Participants in FB+Friends Group: These participants were recruited into the FB+Friends group through week 8 of the intervention
Period: Overall Study
Arm/Group | FB+Friends | FB Only | Non-Randomized Participants in FB+Friends Group
Started | 40 | 40 | 54
Completed | 40 | 39 | 47
Not Completed | 0 | 1 | 7
Not completed — Lost to Follow-up | 0 | 1 | 7

BASELINE CHARACTERISTICS:
Population: Wave 2 Randomized Sample
Groups:
- FB+Friends: FB+Friends is a Facebook-delivered weight loss intervention. For this group, the study team continued to enroll participants through week 8.
  FB + Friends: Participants will receive a weight loss intervention delivered in an online context. The online coaches will post daily content, respond to questions, address concerns, and encourage engagement. The weight loss intervention is based on the Diabetes Prevention Program (DPP), an evidence-based weight loss program focused on lifestyle changes. The goals for the intervention are 175 minutes of moderate physical activity per week and an overall weight loss of 7%. Each participant will get an individualized calorie goal that would facilitate a 1-2 lbs. weight loss weekly. Participants will also be encouraged to use an app such as MyFitnessPal to track daily diet. For this arm, the study team will keep recruitment open for this condition to allow enrollment of new participants through week 8.
- Non-Randomized Participants in FB+Friends Group: This group of participants were enrolled into the FB+Friends group during weeks 1-8 of the intervention, thereby receiving the same intervention as that group.
- Total: Total of all reporting groups
Arm/Group | FB+Friends | FB Only | Non-Randomized Participants in FB+Friends Group | Total
Number analyzed (Participants) | 40 | 40 | 54 | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.0 (10.6) | 40.4 (11.8) | 40.3 (10.6) | 40.2 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 34 | 50 | 118
  Male | 6 | 6 | 4 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4 | 8
  Not Hispanic or Latino | 39 | 36 | 50 | 125
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 3 | 4 | 10
  White | 36 | 36 | 44 | 116
  More than one race | 1 | 0 | 3 | 4
  Unknown or Not Reported | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 54 | 134
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 34.0 (4.6) | 34.8 (5.4) | 34.5 (4.3) | 34.4 (5.0)

OUTCOME MEASURES:

1. Primary Outcome: Engagement
Description: Number of Facebook "likes" and other reactions, replies, posts, and polls per participant during the 16 week program.
Time Frame: 4 months
Population: Wave 2 All Randomized
Measure: Median (Inter-Quartile Range); unit: Total Engagements
Groups:
- FB+Friends: FB+Friends is a Facebook-delivered weight loss intervention. The study team will keep recruitment open for this condition to allow enrollment through week 8.
- FB Only: FB Only Facebook-delivered weight loss intervention including only study participants.
- Non-Randomized Participants in FB+Friends Group: These participants were recruited into the FB+Friends group during weeks 1-8.
Arm/Group | FB+Friends | FB Only | Non-Randomized Participants in FB+Friends Group
Number analyzed (Participants) | 40 | 40 | 54
Total Engagements | 77.00 [29.25 to 271.50] | 116.50 [28.50 to 174.00] | 46.0 [25.75 to 96.25]
Statistical Analysis 1: Comparison: FB+Friends vs FB Only; Mann-Whitney U Test; Test type: Superiority; p = 0.72, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Retention
Description: The number of participants who complete the follow-up assessment in each condition.
Time Frame: 4 months
Population: Wave 2 Only
Measure: Count of Participants; unit: Participants
Groups:
- Non-Randomized Participants in FB+Friends Group: These participants were enrolled into the FB+Friends group between weeks 1-8.
Arm/Group | FB+Friends | FB Only | Non-Randomized Participants in FB+Friends Group
Number analyzed (Participants) | 40 | 40 | 54
Participants | 40 | 39 | 47
Statistical Analysis 1: Comparison: FB+Friends vs FB Only; Chi square test comparing proportion retained in each condition; Test type: Superiority; p = 0.31, Chi-squared

3. Primary Outcome: Number of Participants Rating the Intervention 'Acceptable
Description: Participants will rate acceptability of the online intervention. Acceptability was assessed with a single item during the follow-up survey: "How likely are you to recommend the program to a friend?" (responses on a 5-point Likert scale from not at all likely to very likely). Acceptability was categorized into acceptable, defined as responses of a little bit likely, somewhat likely, likely, and very likely, and unacceptable was defined as response of not at all likely.
Time Frame: 4 months
Population: Wave 2 Participants Who Completed Acceptability Survey Question
Measure: Count of Participants; unit: Participants
Arm/Group | FB+Friends | FB Only | Non-Randomized Participants in FB+Friends Group
Number analyzed (Participants) | 35 | 39 | 47
Participants | 31 | 36 | 44
Statistical Analysis 1: Comparison: FB+Friends vs FB Only; Test type: Superiority; p = 0.69, Chi-squared

4. Secondary Outcome: Percent Weight Loss
Description: We calculated percent weight loss from baseline to 4 months.
Time Frame: Baseline to 4 months
Population: Randomized Sample; FB Only condition excludes 1 participant for pregnancy
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- FB+Friends: FB+Friends is a Facebook-delivered weight loss intervention. For this group, the study team continued to enroll participants through week 8.
- Non-Randomized Participants in FB+Friends Group: These participants were enrolled into the FB+Friends group during weeks 1-8.
Arm/Group | FB+Friends | FB Only | Non-Randomized Participants in FB+Friends Group
Number analyzed (Participants) | 40 | 39 | 51
percent change | -3.0844 (4.28) | -1.8713 (4.41) | -2.8 (4.5)
Statistical Analysis 1: Comparison: FB+Friends vs FB Only; We compared mean percent weight loss from baseline across groups with a one-way ANOVA. One participant became pregnant and thus removed from the analysis. This analysis is exploratory given that this pilot study was not powered to detect weight loss differences between groups; Test type: Superiority; p = 0.218, ANOVA

5. Secondary Outcome: Diet
Description: The percentage of intervention days that a participant tracked diet and/or exercise in MyFitnessPal app. Any entry was counted as a day of tracking.
Time Frame: 4 Months
Population: randomized wave 2 sample
Measure: Mean (Standard Deviation); unit: percentage of days of diet tracking
Groups:
- FB Only: FB Only is a Facebook-delivered weight loss intervention including only study participants.
Arm/Group | FB+Friends | FB Only | Non-Randomized Participants in FB+Friends Group
Number analyzed (Participants) | 40 | 40 | 54
percentage of days of diet tracking | 37.87 (29.49) | 32.41 (31.00) | 30.12 (28.97)
Statistical Analysis 1: Comparison: FB+Friends vs FB Only; Test type: Superiority; p = 0.421, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the period of 16 weeks.
Description: Adverse events were assessed during follow-up as well as documented when participants reported them during the intervention. Pregnancy was only assessed with female participants.
Groups:
- Non-Randomized Participants in FB+Friends Group: Non-Randomized Participants in the FB+Friends Group includes the participants in this condition who enrolled between week 1 and week 8.
  Participants will receive a weight loss intervention delivered in an online context. The online coaches will post daily content, respond to questions, address concerns, and encourage engagement. The weight loss intervention is based on the Diabetes Prevention Program (DPP), an evidence-based weight loss program focused on lifestyle changes. The goals for the intervention are 175 minutes of moderate physical activity per week and an overall weight loss of 7%. Each participant will get an individualized calorie goal that would facilitate a 1-2 lbs. weight loss weekly. Participants will also be encouraged to use an app such as MyFitnessPal to track daily diet. For this arm, the study team will keep recruitment open for this condition to allow enrollment of new participants through week 8.
Arm/Group | FB+Friends | FB Only | Non-Randomized Participants in FB+Friends Group
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/54
Other Adverse Events (participants affected / at risk) | 13/40 | 6/40 | 0/54
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | FB+Friends (N=40) | FB Only (N=40) | Non-Randomized Participants in FB+Friends Group (N=54)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Weight Gain (General disorders) | 0 | 2 | 0 — Pts gained 5% or more of baseline weight during intervention
Had Surgery or Procedure (Surgical and medical procedures) | 4 | 2 | 0
Began Taking Medication Affecting Weight (General disorders) | 2 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0/34 | 1/34 | 0 — Only Assessed in Females
Respiratory Illness (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Gastrointestinal Illness (Gastrointestinal disorders) | 1 | 0 | 0
Losing Vision Due to Genetic Disorder (Congenital, familial and genetic disorders) | 0 | 1 | 0
Binge Eating Disorder (Psychiatric disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-02-03): https://cdn.clinicaltrials.gov/large-docs/80/NCT02656680/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-20): https://cdn.clinicaltrials.gov/large-docs/80/NCT02656680/SAP_002.pdf
  • Informed Consent Form (2019-09-01): https://cdn.clinicaltrials.gov/large-docs/80/NCT02656680/ICF_001.pdf